CLINICAL TRIAL: NCT04269486
Title: Safety Assessment of the Frequently Used Herbal Medicines at Inpatient Setting: a Multicenter, Prospective Observational Study
Brief Title: A Multicenter Observational Study on Safety of the Herbal Medicines at Inpatient Setting
Status: Terminated | Type: Observational
Why Stopped: The funding stopped while participants recruited slowly
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Collaborators: Semyung University (Other); Dongshin Seoul Korean Medicine Hospital (Unknown); CHUNG YEON Korean Medicine Hospital (Unknown); Korean Medicine Hospital of Pusan National University (Other); DongGuk University (Other)
Responsible Party: Principal Investigator, Dal-Seok Oh, OMD, PhD, Principal Investigator, Korea Institute of Oriental Medicine
Other Study IDs: KIOS1901
Record Dates: First submitted 2019-11-26; First posted 2020-02-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Drug Induced Liver Injury; Drug-Induced Kidney Injury; Herbal Medicine Adverse Reaction
Keywords: Safety; Herbal Medicine; Drug Induced Liver Injury; Drug-Induced Kidney Injury; Prospective Observation; Multicenter Study
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver for AST, ALT, ALP, γ-GT, total Bilirubin and mircoRNA-122, GLDH Kidney for sCr, uCr, BUN and NGAL, KIM-1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inpatient participant: Inpatients who signed the informed consent form that she will be observed during the hospitalization period

SUMMARY:
Prospective observations on safety of the herbal medicines regarding liver and kidney injuries at inpatient setting of four sites in South Korea which are located at each quadrant of the country. In a previous study (PMID 28634823), six women presented liver injuries by herbs and similar findings were also reported. That knowledge has been developed to design the observations of females (19-80 ages) at least 2 weeks' hospitalization with weekly routine lab tests to obtain the occurrence of liver or kidney injuries and the profiles on micro biomarkers throughout the hospitalization period, and then, the follow-up test will be conducted in outpatient setting.

DETAILED DESCRIPTION:
Total 500 inpatients will be observed to assess safety of herbal medicines with the balance of 60 to 110 each site. After obtaining the informed consent from patient, blood draw and urine collection are conducted prior to intake of the herbal medicine, blood draw and urine collection are routinely done every week throughout the whole admission period. The primary outcomes are, 1) liver for alanine aminotransferase (ALT), RUCAM (in case of causality assessment when ALT≥3 upper normal limit) and new biomarker, mircoRNA-122 and 2) kidney for urine creatinine, blood urea nitrogen (BUN) and new biomarker, Neutrophil gelatinase-associated lipocalin (NGAL). The secondary outcomes are, 1) liver for aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyltransferase (γ-GT), total bilirubin and new biomarker, glutamate dehydrogenase (GLDH) and 2) kidney for serum creatinine and new biomarker, kidney injury molecule-1 (KIM-1). The follow-up will be done by the study doctors based on their decision on the inpatient after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Female whose age is between 19 and 80
* Inpatient expected to stay at least 2 weeks and to intake herbal medicine
* Who signed voluntarily informed consent.

Exclusion Criteria:

* Who were short of stay for 2 weeks or stopped intaking herbal medicine
* Who had problems physically or mentally by investigator

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female whose age is between 19 and 80
Study Population: The female inpatients who showed their autonomy and voluntarily signed informed consent on the observations thorughout hospitalization period.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Alanine aminotransferase (ALT) (U/L), if ALT >3 upper normal limit, Roussel uclaf casuality assessment method scoring | Activity change from Admission (0 week; ALT) up to discharge (12 weeks; ALT)
  Routine check-up test item and causality assessment on liver functions
Blood urea nitrogen (BUN) (mg/dL) | Activity change from Admission (0 week; BUN) up to discharge (12 weeks; BUN)
  Routine check-up test item on kidney functions

SECONDARY OUTCOMES:
Liver function tests: AST (U/L), ALP (U/L), γ-GT (U/L), total bilirubin (mg/dL). Drug induced-liver injury biomarkers: microRNA-122 (miR122), Glutamate dehydrogenase (GLDH) | Time-dependent Profiles from Admission (0 week), 1 week, 2 weeks, 3 weeks up to discharge (12 weeks)
  Routine check-up test items and newly developed biomarkers on liver functions
Kidney function tests: Urine creatinine (mg/dL), Serum creatinine (mg/dL). Drug induced-kidney injury biomarkers: Neutrophil gelatinase-associated lipocalin, Kidney Injury Molecule-1 | Time-dependent Profiles from Admission (0 week), 1 week, 2 weeks, 3 weeks up to discharge (12 weeks)
  Routine check-up test items and newly developed biomarkers on kidney functions

CONTACTS AND LOCATIONS:
Overall Officials: Dal-Seok Oh, OMD, PhD, Principal Investigator — Korea Institute of Oriental Medicine
Locations (1):
- Five tertiary Korean Medicine Hospital (Jecheon, Yangsan, Gwangju, Seoul, Bundang), Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Online source on the previous study paper — https://www.ncbi.nlm.nih.gov/pubmed/28634823